CLINICAL TRIAL: NCT06862999
Title: Comparing the Effectiveness of Non-financial Incentive to Participate in a Smartphone Experience Sampling Method Well-being Study: Protocol for a Randomised Controlled Trial
Brief Title: Willingness to Participate in a Daily Smartphone Well-being Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Principal Investigator, Abdur-Rahman, Principal Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-17042-30162
Record Dates: First submitted 2025-03-05; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Willingness to Participate
Keywords: Experience Sampling Method; Willingness to Participate; Neighbourhood studies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Placebo Comparator): Participants in this group will receive no incentive for participating in the future experience sampling study.
  Interventions: Behavioral: No Incentive Email
- Financial Incentive Group (Experimental): Participants in this group will receive a financial incentive for participating in the future experience sampling study.
  Interventions: Behavioral: Financial Incentive Email
- Non-Financial Incentive Group (Experimental): Participants in this group will receive a non-financial incentive for participating in the future experience sampling study.
  Interventions: Behavioral: Social Incentive Email

INTERVENTIONS:
Behavioral: No Incentive Email — Participant will receive an email describing a hypothetical experience sampling study that will happen in King's Cross where he or she is an inhabitant as a worker, resident, or visitor. However, this email will not include any promised compensation for future participation in the hypothetical wellbeing study in the neighbourhood. This group serves as the control group to compare the effects of incentives on participation rates.
  Arms: Control Group
Behavioral: Financial Incentive Email — Participant will receive an email describing a hypothetical experience sampling study that will happen in King's Cross where he or she is an inhabitant as a worker, resident, or visitor. This email will include a paragraph that describes a compensation for participation in the future study. The type of compensation that will be offered is a financial compensation, which is a chance of enter a prize draw to win a 4 X £100 voucher which can be used to purchase goods and services within the King's Cross neighbourhood in London.
  Arms: Financial Incentive Group
Behavioral: Social Incentive Email — Participant will receive an email describing a hypothetical experience sampling study that will happen in King's Cross where he or she is an inhabitant as a worker, resident, or visitor. This email will include a paragraph that describes a compensation for participation in the future study. The type of compensation that will be offered is a non-financial compensation, which is an invitation to participate in a social event that will be organised by the researchers and the neighbourhood asset manager team at the end of the research project. This event will be exclusive and it will be an opportunity for participants to socialize with other study participants in the neighbourhood. It will also be an opportunity for the study participants to feel they are contributing a change to the neighbourhood and will be able to articulate their views about the wellbeing research findings which is expected to be used to inform future interventions in the neighbourhood.
  Arms: Non-Financial Incentive Group

SUMMARY:
This clinical trial aims to compare the effectiveness of financial and social incentives in motivating urban populations to participate in Experience Sampling Method (ESM) wellbeing studies and explore alternative incentive preferences to increase participation.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the comparison of two incentives to determine their effectiveness for motivating an urban population to participate in a Experience Sampling Method wellbeing studies. It will also investigate alternative incentive preferences that can motivate the population. The main questions it aims to answer are:

* Does the provision of a financial incentive or social incentive to neighbourhood research participants increase the willingness of individuals to participate in ESM research compared to offering no incentive?
* What are the reasons for unwillingness to participate in ESM studies?
* What are the alternative incentive preference that could increase willingness to participate in ESM studies?

Researchers will compare monetary incentive (4 x £100 prize draw qualification) to a non-monetary incentive (invitation to end of project social event to engage research findings) to how they influence willingness to participate compared to offering no incentive.

Participants will:

* Receive receive an email describing a future experience sampling study in the neighbourhood for at least two times.
* Complete a survey to indicate their positive or negative interest in the hypothetical study.

ELIGIBILITY:
Inclusion Criteria:

* Registered on the King's Cross community smartphone application.
* App users living, working, or have previously visited King's Cross
* Given consent to receive email communications during their smartphone app sign-up.

Exclusion Criteria:

* Users of the King's Cross community smartphone app who have not given consent to receive email communication about the neighbourhood

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Willingness to participate | From enrollment to the end of treatment at 7 weeks
  Measure the proportion of participants in each arm who agree to participate in the experience sampling study.

OTHER OUTCOMES:
Reasons for non-participation | From enrollment to the end of treatment at 7 weeks
  Participants who are not willing to participate in the future experience sampling study will be asked to indicate four out of seven reasons for the unwillingness.
Alternative Incentive Preferences | From enrollment to the end of treatment at 7 weeks
  Participants who are not willing to participate in the future experience sampling study and who select "inadequate compensation" as one of the reasons for not participating will be asked to select desired incentives from a list of seven options that could motivate a change in participation decision.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley-Anne Carter, Principal Investigator — University of Manchester; Jack Benton, Principal Investigator — University of Manchester; Jamie Anderson, Principal Investigator — University of Manchester
Locations (1):
- Related Argent, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
With the exception of the identifying email addresses, the demographic and outcome data that was collected from the participant will be publicly made available on UK Data Service ReShare, a platform for archiving research data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication and the duration the data will be made accessible for is based on the terms and conditions attached to the ReShare platform where the data will be archived.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research